CLINICAL TRIAL: NCT02899793
Title: A Phase II Evaluation of Pembrolizumab, a Humanized Antibody Against PD-1, in the Treatment of Persistent or Recurrent Hypermutated/Ultramutated Endometrial Cancer Identified by Next Generation Sequencing (NGS) and Comprehensive Genomic Profiling (CGP)
Brief Title: Pembrolizumab in Ultramutated and Hypermutated Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1605017712; 000 (Other: CTGTY)
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab 200 mg, Q3W, IV Infusion, Day 1 of each 3 week cycle
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg (fixed dose) IV every 3 weeks (+/- 3 days) until progression or adverse effects prohibit therapy
  Other Names: MK-3475

SUMMARY:
Primary Objectives: To assess the antitumor activity (proportion of objective response by RECIST 1.1 criteria) of pembrolizumab with objective tumor response in patients with persistent, recurrent or metastatic endometrial cancer harboring an ultra-mutated or hyper-mutated (MMR gene-defective) phenotype identified by next generation sequencing (NGS) and comprehensive genomic profiling (CGP). To determine the nature and degree of toxicity of pembrolizumab as assessed by CTCAE in patients with persistent, recurrent or metastatic endometrial carcinoma. Secondary Objective(s): To estimate the duration of progression-free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed endometrial cancer that is recurrent or progressive following at least one prior chemotherapy regimen.
2. Patients with the following histologic epithelial cell types are eligible: Endometrioid adenocarcinoma, serous adenocarcinoma, clear cell carcinoma, undifferentiated carcinoma, mixed epithelial carcinoma, carcinosarcoma, and adenocarcinoma not otherwise specified (N.O.S.).
3. Tumors must demonstrate ultramutation (POLE/POLD1-mutation) and/or hyper-mutation (due to MMR gene defect) in a representative primary or metastatic tumor site by next generation sequencing (NGS) and Comprehensive Genomic Profiling (CGP) testing, and/or standard PCR-based DNA microsatellite instability (MSI) and immunohistochemistry (IHC).
4. All patients must have measurable disease by RECIST 1.1.
5. Patients must have a ECOG performance status of 0 or 1.
6. Women of childbearing potential must have a negative urine and serum pregnancy test within 72 hours prior to receiving first dose and must be willing to use contraceptive through 120 days of last dose of Pembrolizumab.
7. Patients must have recovered from effects of recent surgery, radiotherapy, or chemotherapy. Patients with ≥ Grade 2 neuropathy are eligible.
8. Patients may have received prior radiation therapy for treatment of endometrial cancer. Prior radiation therapy may have included pelvic radiation therapy, extended field pelvic/para-aortic radiation therapy, intravaginal brachytherapy and/or palliative radiation therapy. All radiation therapy must be completed at least 4 weeks prior to the first date of study therapy.
9. Patients may have received prior hormonal therapy for treatment of endometrial carcinoma. All hormonal therapy must be discontinued at least one week prior to the first date of study therapy.
10. Patients may have received prior therapy (including chemotherapy, biologic/targeted therapy and immunotherapy) for treatment of endometrial cancer. All therapy must be discontinued at least 3 weeks prior to the first date of study therapy. Any investigational agent must be discontinued at least 30 days prior to the first date of study therapy.
11. Chemotherapy administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a systemic chemotherapy regimen.
12. Patients are allowed to receive, but not required to receive, up to 4 additional lines of therapy.
13. At least 4 weeks must have elapsed since the patient underwent any major surgery (e.g., major: laparotomy, laparoscopy) There is no delay in treatment for minor procedures (e.g., tumor FNA or core biopsy, venous access device placement).
14. Have demonstrated adequate organ function. All screen labs should be performed within 14 days of treatment initiation
15. Patients must have signed an approved informed consent and authorization permitting release of personal health information.
16. Patients must be 18 years or older

Exclusion Criteria:

1. Patients who have had prior therapy with nivolumab, pembrolizumab or with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune check point pathways.
2. History of severe hypersensitivity reaction to any monoclonal antibody.
3. Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure and unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Patients who are pregnant or nursing. The effects of pembrolizumab on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. WOCBP should use an adequate method to avoid pregnancy for 23 weeks after the last dose of investigational drug. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IV/L or equivalent units of HCG) within 24 hours prior to the start of pembrolizumab. Women must not be breastfeeding.
5. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile or have undergone definitive radiation) do not require contraception.
6. Patients with known brain metastases or leptomeningeal metastases are excluded unless the following conditions are met: Metastases have been treated and there is no evidence of progression by CT scan or magnetic resonance imaging (MRI) prior to the first dose of pembrolizumab administration). There must also be no requirement for immunosuppressive doses of systemic corticosteroids (>10 mg/day prednisone equivalents) for at least 1 week prior to study drug administration.
7. Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). Patients should be excluded if they have a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection (e.g., HCV RNA [qualitative] is detected).
8. Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as SLE, connective tissue diseases, scleroderma, inflammatory bowel disease (IRB), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patient with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.

   NOTE: Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event).
9. Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if <10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
10. Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, abdominal/pelvic fistula, gastrointestinal perforation, GI obstruction and/or who require parenteral hydration and/or nutrition..
11. Has a known history of active TB (Bacillus Tuberculosis)
12. Hypersensitivity to pembrolizumab or any of its excipients.
13. Prior invasive malignancy (except non-melanomatous skin cancer such as basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer) unless disease free for a minimum of 3 years.
14. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
15. Has an active infection requiring intravenous systemic therapy.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Has not recovered from adverse events to <Grade 1 or prior treatment level due to a previously administered agent. Subjects with Grade <2 neuropathy or alopecia of any grade are an exception to this criterion and may qualify for the study.
19. Has a known additional malignancy that progressed or required active treatment within the last five years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
20. Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
21. Patients should not have used investigational agents or device within 4 weeks prior to first dose.
22. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro D. Santin, M.D, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ettorre VM, Bellone S, Greenman M, McNamara B, Palmieri L, Sethi N, Demirkiran C, Papatla K, Kailasam A, Siegel ER, Ratner E, Santin AD. A phase 2 trial of pembrolizumab for recurrent Lynch-like versus sporadic endometrial cancers with microsatellite instability (NCT02899793): Updated survival and response analyses. Gynecol Oncol. 2025 Jun;197:110-115. doi: 10.1016/j.ygyno.2025.04.591. Epub 2025 May 6. PMID 40334308
- [Derived] Bellone S, Roque DM, Siegel ER, Buza N, Hui P, Bonazzoli E, Guglielmi A, Zammataro L, Nagarkatti N, Zaidi S, Lee J, Silasi DA, Huang GS, Andikyan V, Damast S, Clark M, Azodi M, Schwartz PE, Tymon-Rosario JR, Harold JA, Mauricio D, Zeybek B, Menderes G, Altwerger G, Ratner E, Alexandrov LB, Iwasaki A, Kong Y, Song E, Dong W, Elvin JA, Choi J, Santin AD. A phase 2 evaluation of pembrolizumab for recurrent Lynch-like versus sporadic endometrial cancers with microsatellite instability. Cancer. 2022 Mar 15;128(6):1206-1218. doi: 10.1002/cncr.34025. Epub 2021 Dec 7. PMID 34875107
- [Derived] Bellone S, Roque DM, Siegel ER, Buza N, Hui P, Bonazzoli E, Guglielmi A, Zammataro L, Nagarkatti N, Zaidi S, Lee J, Silasi DA, Huang GS, Andikyan V, Damast S, Clark M, Azodi M, Schwartz PE, Tymon-Rosario J, Harold J, Mauricio D, Zeybek B, Menderes G, Altwerger G, Ratner E, Alexandrov LB, Iwasaki A, Kong Y, Song E, Dong W, Elvin J, Choi J, Santin AD. A phase II evaluation of pembrolizumab in recurrent microsatellite instability-high (MSI-H) endometrial cancer patients with Lynch-like versus MLH-1 methylated characteristics (NCT02899793). Ann Oncol. 2021 Aug;32(8):1045-1046. doi: 10.1016/j.annonc.2021.04.013. Epub 2021 Apr 28. No abstract available. PMID 33932502

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 25
Excluded From Analysis Due to Tumor Status | 1
Completed | 24
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Characteristic data presented here is from the 24 participants that completed
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
International Federation of Gynecology and Obstetrics (FIGO) Stage at diagnosis, No. (%) [Count of Participants; unit: Participants] — Stage I: The cancer is limited to the organ of origin. Stage II: The cancer has spread to nearby tissues or organs. Stage III: The cancer has spread to distant lymph nodes or tissue within the pelvis. Stage IV: The cancer has spread to distant sites (metastasis).
  Participants
    Stage I | 12
    Stage II | 1
    Stage III | 8
    Stage IV | 3
Histology/grade of Endometrial Adenocarcinoma (EAC) [Count of Participants; unit: Participants] — G1: The cells are well differentiated. (Low grade tumor), G2: The cells are moderately differentiated., G3: The cells are poorly differentiated. (High grade tumor)
  Participants
    EAC G1 | 2
    EAC G2 | 9
    EAC G3 | 13
Microsatellite instability-high (MSI-H)/mismatch repair deficiency (dMMR) Subgroups Characteristics [Count of Participants; unit: Participants]
  Lynch-like | 6
  Methylated | 18

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Objective Tumor Response as Assessed by RECIST 1.1- Overall Response Rate (ORR)
Description: RECIST (Response Evaluation Criteria In Solid Tumors) is a set of published rules that define when cancer patients improve ("respond"), stay the same ("stable") or worsen ("progression") during treatments. Complete Response (CR) = complete disappearance of all clinical evidence of disease; Partial Response (PR) = regression of measurable disease; Stable Disease (SD) = failure to attain CR, PR, or PD; Progressive Disease (PD) = PD in any compartment; Relapse = recurrence of disease in prior CR in any compartment.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 24
Participants
  CR | 5
  PR | 9
  SD | 7
  PD | 3
Statistical Analysis 1: Comparison: Pembrolizumab; Subgroup difference in ORRs; Test type: Superiority; p = 0.024, Fisher Exact

2. Primary Outcome: Toxicity Grade of Adverse Events as Assessed by CTCAE v4
Description: Common Terminology Criteria for Adverse Events (CTCAE) are a set of criteria for the standardized classification of adverse effects of drugs used in cancer therapy. Number of patients affected by each adverse event grade for Other (non-serious) adverse events with in the treatment period.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 25
Participants
  Grade 1 | 19
  Grade 2 | 6
  Grade 3 | 0
  Grade 4 | 0

3. Secondary Outcome: Duration of Progression-free Survival (PFS)
Description: Progression-free survival is defined as the duration of time from study entry to time of progression, death, or the date of last contact, whichever occurs first.
Time Frame: 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 24
months | 27.4 [10.7 to NA] — Upper limit confidence interval was not reached due to insufficient number of events

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 24
months | 71.5 [28.6 to NA] — Upper limit confidence interval was not reached due to insufficient number of events

ADVERSE EVENTS:
Time Frame: 6 years
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 12/25
Serious Adverse Events (participants affected / at risk) | 23/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=25)
Hyperthyroidism (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Fever (General disorders) | 2
Pain (General disorders) | 1
Urinary tract infection (Infections and infestations) | 4
Ankle fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=25)
Fatigue (General disorders) | 16
Pain (General disorders) | 10
Edema limbs (General disorders) | 8
Fever (General disorders) | 3
Chills (General disorders) | 2
Infusion related reaction (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 3
Musculoskeletal and connective tissue disorder -Other, specify (Musculoskeletal and connective tissue disorders) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Urinary tract infection (Infections and infestations) | 8
Infections and infestations - Other, specify (Infections and infestations) | 5
Upper respiratory infection (Infections and infestations) | 5
Skin infection (Infections and infestations) | 3
Tooth infection (Infections and infestations) | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Hematuria (Renal and urinary disorders) | 4
Urinary frequency (Renal and urinary disorders) | 4
Urinary incontinence (Renal and urinary disorders) | 3
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Hypothyroidism (Endocrine disorders) | 6
Endocrine disorders - Other, specify (Endocrine disorders) | 2
Creatinine increased (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Weight loss (Investigations) | 2
Headache (Nervous system disorders) | 4
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 2
Anemia (Blood and lymphatic system disorders) | 4
Atrial fibrillation (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 2
Dry eye (Eye disorders) | 3
Eye disorders - Other, specify (Eye disorders) | 2
Anxiety (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT02899793/Prot_SAP_000.pdf